CLINICAL TRIAL: NCT01059149
Title: Safety and Long-term Effectiveness of High Frequency Repetitive Transcranial Magnetic Stimulation at the Subacute Phase of Ischaemic Stroke
Brief Title: Safety and Long-term Effectiveness of High Frequency Repetitive Transcranial Magnetic Stimulation of Stroke (RAICup)
Acronym: RAICup
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P080604
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2012-11

CONDITIONS: Nervous System Diseases; Stroke; Cerebrovascular Disorders; Brain Infarction; Brain Ischemia
Keywords: Rehabilitation; Transcranial magnetic stimulation; Brain magnetic stimulation; Repetitive; Stroke; Subacute
MeSH Terms: conditions — Nervous System Diseases; Stroke; Cerebrovascular Disorders; Brain Infarction; Brain Ischemia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- receive real rTMS (Experimental): For real rTMS, pulses will be delivered at a frequency of 5 Hz for 6s with a 54s interval, with an intensity equal of 90% of the motor threshold as established at Baseline. 20-min real stimulation sessions will be administered 5 days a week for a period of 2 weeks
  Interventions: Device: repetitive transcranial magnetic stimulation
- sham rTMS (Placebo Comparator): For sham rTMS, procedures will be identical to those used for real rTMS with the exception that a placebo procedures will be used administered 5 days a week for a period of 2 weeks.
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — MagPro x100 (MagVenture A/S, DANEMARK)

SUMMARY:
The aim of the study is to determine if 2-week repetitive transcranial magnetic stimulation at the subacute phase of stroke (between day 7 and day 14) improves significantly arm motility at 3 months with remaining effect at one year, without significant adverse effect.

DETAILED DESCRIPTION:
Stroke survivors may be left with disability involving speech or residual arm or leg weakness. Despite spontaneous improvement on the weeks following stroke, the importance of final disability is unpredictable. If the core of the infarct is represented by dead neurons, the neurons from adjacent areas seem to be staggered and their lack of excitability has been correlated to a bad prognosis. Repetitive transcranial magnetic stimulation (rTMS) seems to be a promising technique since high frequency rTMS can increase excitability of the targeted neurons.

The aim of the study is to evaluate after 2 weeks of 20 min of rTMS each day: 1) the improvement of arm function and neurological and disability scales, immediately after the 2-week session, at one month, 3 months and evaluate the remnant effect at 12 months, 2) to correlate these scales to physiological parameters in order to assess the clinical modifications to the electrophysiological modifications, 3) to assert the safety of high frequency rTMS at the subacute phase of ischaemic stroke.

ELIGIBILITY:
Inclusion Criteria:

Single mono hemispheric subcortical and/or cortical ischaemic stroke (documented by CT or MRI) 7 to 21 days before, with moderate arm paresis as defined by a Rankin score <= 4 or not at 4 (in paragraph 5 of NIHSS), in the territory of middle cerebral artery Patients between 18 and 80 years old

Exclusion Criteria:

severe peripheral neuropathy pace-maker, implanted medical pump, metal plate, metal object in the skull or eye History of previous stroke, epileptic seizures, craniotomy, brain trauma Score Rankin > 4 and arm deficit at 4 (paragraph 5 of NIHSS) Score Rankin <=1 Cortical stroke Alertness problems at the time of inclusion Disability previous to stroke Stenosis of internal carotid artery with surgery foreseen within 3 months Uncontrolled medical problem Not able to give informed consent Pregnant or breast-feeding woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Improvement in the arm function in patients treated with rTMS as measured by the ARA (Action Research Arm) test at 3 months follow-up compared to the sham treated patients | 3 months

SECONDARY OUTCOMES:
Improvement of hand function as measured by ARA test and Box and Block test at 2-week, 1 month, 3 months and 1 year follow-up | 1 year
Improvement of neurological score (NIHSS), disability scales (Barthel, Rankin), spasticity scales (Ashworth) | 1 year
Identify groups of good and bad responders in correlation to other excitability parameters and other parameters known to impede functional outcome (importance of the initial deficit, infarct volume, lesion on the CORTICO-spinal tract) | 1 year
Period before the patient is able to go back home | 1 year
Influence of the side of the stimulation on depression (Hamilton scale) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: KUBIS Nathalie, MD, PhD, Principal Investigator — Physiology Department, Hôpital Lariboisière, Paris
Locations (1):
- Physiology Department, Hôpital Lariboisière, Université Paris 7, Paris, Île-de-France Region, France